CLINICAL TRIAL: NCT01055821
Title: A Phase II Randomized, Multicenter, Open-label Study of TG4040 (MVA-HCV) in Combination With Pegylated Interferon Alfa-2a and Ribavirin Versus Pegylated Interferon Alfa-2a and Ribavirin in Treatment-naïve Patients With Chronic Genotype 1 Hepatitis C.
Brief Title: Efficacy of the Therapeutic Vaccine TG4040 Combined With Pegylated Interferon and Ribavirin in Chronic HCV Patients
Acronym: HCVac
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Transgene (Industry)
Responsible Party: G Honnet, Transgene
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TG4040.02
Record Dates: First submitted 2010-01-21; First posted 2010-01-26 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Chronic Hepatitis C Infection
Keywords: Hepatitis C; Vaccine; HCVac; MVA-HCV
MeSH Terms: conditions — Hepatitis C | interventions — Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A (Active Comparator): Standard of care (SOC)
  Interventions: Drug: pegylated interferon and ribavirin
- Arm B (Experimental): Vaccine and Standard of care
  Interventions: Biological: TG4040 + SOC
- Arm C (Experimental): vaccine and standard of care
  Interventions: Biological: TG4040 + SOC

INTERVENTIONS:
Drug: pegylated interferon and ribavirin — 48 weeks
  Arms: Arm A
Biological: TG4040 + SOC — 6 injections
  Arms: Arm B
Biological: TG4040 + SOC — 13 injections
  Arms: Arm C

SUMMARY:
The primary objective of this protocol is to study the effect of the standard of care in hepatitis C (pegylated interferon and ribavirin) associated with therapeutic vaccine TG4040 on the viral load of treatment-naïve patients with chronic genotype 1 hepatitis C infection.

ELIGIBILITY:
Inclusion Criteria:

* Chronically infected patients with Hepatitis C virus Genotype 1 (1a or 1b) with detectable viremia (HCV RNA in blood) for more than 6 months and naïve to treatment;
* Patients must have compensated liver disease, with no history of ascites, jaundice, hepatic encephalopathy or bleeding from esophageal or gastric varices requiring beta-blockers;
* No histological evidence of hepatic cirrhosis (including compensated cirrhosis) based on a liver biopsy taken within 24 months prior to baseline; or on a FibroScan® performed within 6 months prior to treatment which indicates the absence of liver cirrhosis, i.e., stage < F4 (METAVIR); in case of no available results, a liver biopsy will be performed prior to treatment;
* All laboratory parameters must be grade 0 or 1 (as per CTCAE criteria) except for alanine amino-transferase (ALT), aspartate amino-transferase (AST), gamma glutamyl transferase (GGT) and alkaline phosphatase (ALP) for which a grade 2 will be allowed if stated non clinically significant;
* No co-infection with Human Immunodeficiency Virus (HIV) or hepatitis B virus (HBsAg positive);
* No intravenous (IV) drug or alcohol abuse;
* Serum thyroid stimulating hormone (TSH) levels within normal ranges, regardless of treatment with L-thyroxin;
* Normal electrocardiogram (ECG);
* Normal retinal examination (eye fundus) within last 12 months for diabetic patients or patients suffering from high blood pressure;
* Negative pregnancy test in women of childbearing potential (a woman who is two years post-menopausal or surgically sterile is not considered to be of childbearing potential);
* Female patients and female partners of male patients (if childbearing potency) must agree to use two effective methods of birth control during the study and for 6 months after the end of treatment. One of the methods needs to be a 'barrier' method (condom or diaphragm);

Exclusion Criteria:

* Prior treatment for hepatitis C;
* Malignancy within the last 5 years; except for patients with history of squamous cell skin cancer or basal cell skin cancer who will be enrolled, unless patients have a history of skin cancer at the vaccination site;
* Diagnosed or suspected hepatocellular carcinoma;
* History of psychiatric conditions including, but not limited to, psychosis, suicidal ideations, or major depression. Patients with mild to moderate depression in the past and no prior history of suicidal gestures or attempts may be enrolled if, in the Investigator's opinion, they are suitable for treatment;
* Serious, concomitant medical disorder, including active systemic infection and proven or suspected immunosuppressive disorder;
* History of immunodeficiency or autoimmune disease including autoimmune hepatitis, allogenic transplant, or pre-existing autoimmune or antibody-mediated disease including, but not limited to: systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjogren's syndrome, or autoimmune thrombocytopenia;
* Administration of any vaccine or immunoglobulin within 30 days before the first dose of TG4040 /SOC;
* Significant cardiovascular disease (e.g., New York Heart Association [NYHA] class 3 congestive heart failure; myocardial infarction within the past 6 months; unstable angina; coronary angioplasty within the past 6 months; or uncontrolled arterial or ventricular cardiac arrhythmias);
* Systemic corticosteroid therapy or other immunosuppressive/immunomodulating drugs (e.g. Cyclosporine) within 2 months prior to first TG4040/SOC administration; corticosteroid nasal sprays, inhaled steroids for asthma and/or topical steroids are allowed;
* Any known allergy to interferon (IFN), RBV and/or their excipients;
* Any medical contraindications to IFN and/or RBV;
* Any known allergy to eggs;
* Women who are breastfeeding;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2010-05; Primary Completion 2012-10 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
complete early virologic response | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital, Hanover, Germany

REFERENCES:
- [Derived] Di Bisceglie AM, Janczweska-Kazek E, Habersetzer F, Mazur W, Stanciu C, Carreno V, Tanasescu C, Flisiak R, Romero-Gomez M, Fich A, Bataille V, Toh ML, Hennequi M, Zerr P, Honnet G, Inchauspe G, Agathon D, Limacher JM, Wedemeyer H. Efficacy of immunotherapy with TG4040, peg-interferon, and ribavirin in a Phase 2 study of patients with chronic HCV infection. Gastroenterology. 2014 Jul;147(1):119-131.e3. doi: 10.1053/j.gastro.2014.03.007. Epub 2014 Mar 18. PMID 24657484